CLINICAL TRIAL: NCT03028220
Title: Impact on Hypoglycaemia Awareness of Real Time CGM and Intermittent Continuous
Brief Title: Impact on Hypoglycaemia Awareness of Real Time CGM and Intermittent Continuous Glucose Data
Acronym: IHART-CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15HH2875
Record Dates: First submitted 2016-12-16; First posted 2017-01-23 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia; Impaired Awareness of Hypoglycemia; Type1diabetes
Keywords: Type 1 Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real time continuous glucose monitoring (Active Comparator): Use of Dexcom G5 continuous glucose monitoring
  Interventions: Device: Dexcom G5 Continuous Glucose Monitor
- Flash glucose monitoring (Active Comparator): Use of Abbott FreeStyle Libre flash glucose monitoring
  Interventions: Device: Abbott Freestyle Libre

INTERVENTIONS:
Device: Dexcom G5 Continuous Glucose Monitor — Real time continuous glucose sensor connected to monitor providing data and alarms and alerts for glucose trends and values
  Arms: Real time continuous glucose monitoring
Device: Abbott Freestyle Libre — Continuous glucose recording device which reports glucose concentration and trend on demand, along with a retrospective review of the last 8 hours glucose data
  Arms: Flash glucose monitoring

SUMMARY:
This clinical study proposes to assess the impact of Libre on frequency, duration and severity of hypoglycaemia, compared with the Dexcom G5 realtime CGM and will focus on people with impaired awareness of hypoglycaemia.

DETAILED DESCRIPTION:
Good glucose control in type 1 diabetes is associated with a reduced risk of diabetes complications and self monitoring of glucose levels is an important component of achieving and maintaining glucose control. Continuous glucose monitoring (CGM) improves overall glucose control in all age groups when used continuously, and reduces the incidence of low blood glucose (hypoglycaemia) in people with good glucose control. Hypoglycaemia is one of the commonest metabolic complications of type 1 diabetes and, if it occurs frequently, people can become less aware of it. This reduced aware of hypoglycaemia has significant risks including seizures, coma and even death, and has an impact on people's ability to drive and function.

The Abbott Libre intermittent glucose monitoring system provides up to 8 hours of retrospective continuous glucose monitoring data to users when the monitor is waved in proximity with the sensor. In contrast to realtime CGM the Libre system sensor is used for 14 days and is non-adjunctive (does not require calibration to capillary blood glucose).

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Type 1 diabetes confirmed on the basis of clinical features and a fasting c-peptide <200 pmol/L
* Severe hypoglycaemic event in the last 12 months requiring third party assistance OR a Gold Score ≥ 4
* Type 1 diabetes for greater than 3 years
* On an intensified multiple dose insulin injection regimen for > 6 months (MDI)
* Previous type 1 diabetes structured education (either group or 1:1)

Exclusion Criteria:

* Use of CGM or Libre device within the last 6 months (except short periods of diagnostic blinded use under clinic supervision)
* Use of regular paracetamol
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials, except at the discretion of the chief investigator
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Unable to participate due to other factors, as assessed by the Chief Investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, FRCP, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avari P, Moscardo V, Jugnee N, Oliver N, Reddy M. Glycemic Variability and Hypoglycemic Excursions With Continuous Glucose Monitoring Compared to Intermittently Scanned Continuous Glucose Monitoring in Adults With Highest Risk Type 1 Diabetes. J Diabetes Sci Technol. 2020 May;14(3):567-574. doi: 10.1177/1932296819867688. Epub 2019 Aug 2. PMID 31375042
- [Derived] Reddy M, Jugnee N, El Laboudi A, Spanudakis E, Anantharaja S, Oliver N. A randomized controlled pilot study of continuous glucose monitoring and flash glucose monitoring in people with Type 1 diabetes and impaired awareness of hypoglycaemia. Diabet Med. 2018 Apr;35(4):483-490. doi: 10.1111/dme.13561. Epub 2017 Dec 29. PMID 29230878

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant in the CGM group was randomised and completed the trial but the CGM data could not be analysed due to an uploading error. All other data was analysed for this participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.5 [45 to 64.5] | 48.5 [34 to 63] | 49.5 [37.5 to 63.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 12 | 12 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: % Time Spent in Hypoglycaemia (<3.3mmol/L, 60mg/dL)
Description: Percentage time spent in hypoglycaemia (<3.3mmol/L, 60mg/dL) change from baseline
Time Frame: 10 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time <3.3mmol/l
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percentage of time <3.3mmol/l | -3.0 [-5.0 to -0.3] | 1.3 [-1.4 to 3.6]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: % Time Spent in Hypoglycaemia (<2.8mmol/L, 50mg/dL)
Description: Percentage time spent in hypoglycaemia (<2.8mmol/L, 50mg/dL) change from baseline
Time Frame: 10 weeks
Measure: Median (95% Confidence Interval); unit: percentage of time <2.8mmol/l
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percentage of time <2.8mmol/l | -1.2 [-4.3 to -0.5] | 1.3 [-1.0 to 2.4]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: % Time Spent in Hypoglycaemia (<3.9mmol/L, 70mg/dL)
Description: Percentage time spent in hypoglycaemia (<3.9mmol/L, 70mg/dL) change in baseline to endpint
Time Frame: 10 weeks
Measure: Median (95% Confidence Interval); unit: percentage of time <3.9mmol/l
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percentage of time <3.9mmol/l | -2.7 [-6.1 to -0.1] | 0.6 [-2.1 to 5.4]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: % Time Spent in Euglycaemia (3.9-7.8mmol/L, 70-140mg/dL)
Description: Percentage time spent in euglycaemia (3.9-7.8mmol/L, 70-140mg/dL) change in baseline to endpoint
Time Frame: 10 weeks
Measure: Median (95% Confidence Interval); unit: percentage of time >3.9<7.8 mmol/l
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percentage of time >3.9<7.8 mmol/l | 10.6 [3.3 to 14.4] | 5.9 [-2.4 to 9.0]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 1.00, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: % Time Spent in Euglycaemia (3.9-10mmol/L, 70-180mg/dL)
Description: Percentage time spent in euglycaemia (3.9-10mmol/L, 70-180mg/dL) change in baseline to endpoint
Time Frame: 10 weeks
Measure: Median (95% Confidence Interval); unit: percentage of time >3.9<10 mmol/l
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percentage of time >3.9<10 mmol/l | 12.7 [7.2 to 15.8] | 5.3 [1.1 to 11.7]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 1, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: % Time Spent in Hyperglycaemia (>10mmol/L, 180mg/dL)
Description: Percentage time spent in hyperglycaemia (>10mmol/L, 180mg/dL) change in baseline to endpoint
Time Frame: 10 weeks
Measure: Median (95% Confidence Interval); unit: percentage of time >10mmol/L
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percentage of time >10mmol/L | -8.6 [-13.0 to -1.1] | -7.0 [-16.9 to 1.7]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 0.820, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: % Time Spent in Hyperglycaemia (>15mmol/L, 270mg/dL)
Description: % time spent in hyperglycaemia (>15mmol/L, 270mg/dL) change in baseline to endpoint
Time Frame: 10 weeks
Measure: Median (95% Confidence Interval); unit: percentage of time >15 mmol/l
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percentage of time >15 mmol/l | -4.9 [-8.6 to -0.7] | -3.1 [-5.3 to -0.4]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 0.820, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Hypoglycemia
Description: Number of participants with hypoglycemic excursions
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 0.570, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Severe Hypoglycaemia
Description: Number of participants with episodes of severe hypoglycaemia
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Changes in Glucose Variability Measured
Description: Glucose Variability measured by Coefficient of variation (CV), on a decimal scale of 0-1
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
percent | -0.1 [-0.1 to 0.0] | 0.0 [-0.1 to 0.0]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 0.910, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Glucose Variability Measured by MAGE
Description: Glucose Variability measured by Mean amplitude of Glycaemic Excursions (MAGE)
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
mmol/L | -1.5 [-2.9 to -0.5] | -0.4 [-1.6 to 0.1]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 0.460, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Glucose Variability Measured by CONGA
Description: Glucose Variability measured by Continuous Overlapping Net Glycaemic Action (CONGA)
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: mmol/l
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
Number analyzed (Participants) | 19 | 20
mmol/l | 0.1 [-0.5 to 0.2] | 0.1 [-0.1 to 0.2]
Statistical Analysis 1: Comparison: Real Time Continuous Glucose Monitoring vs Flash Glucose Monitoring; Test type: Other; p = 0.191, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Real Time Continuous Glucose Monitoring | Flash Glucose Monitoring
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03028220/Prot_SAP_000.pdf